CLINICAL TRIAL: NCT04418297
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential, Phase I Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CT-G20 in Subjects With Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CT-G20 in Subjects With Obstructive Hypertrophic Cardiomyopathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The termination criteria of the protocol was met during dose escalation
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-G20 1.2
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-08

CONDITIONS: Cardiomyopathy, Hypertrophic Obstructive
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-G20 (Experimental)
  Interventions: Drug: CT-G20
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT-G20 — oral tablet
  Arms: CT-G20
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, sequential, 5-day treatment, ascending dose study in subjects with obstructive HCM aged 18-70 years. The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of CT-G20.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 70 years, inclusive at Screening
2. Has established diagnosis of HCM defined by standard criteria as a maximal left ventricular wall thickness ≥15 mm at initial diagnosis in the absence of other causative loading abnormalities capable of producing the magnitude of hypertrophy observed or ≥13 mm if the subject has a family history of HCM
3. Has LVOT gradient ≥30 mmHg at rest or LVOT gradient ≥50 mmHg with Valsalva maneuver, due to SAM

Exclusion Criteria:

1. Known infiltrative, genetic or storage disorder causing cardiac hypertrophy that mimics HCM, such as Fabry disease, amyloidosis or Noonan syndrome with LV hypertrophy
2. History of persistent atrial fibrillation prior to Screening or Baseline
3. History of paroxysmal atrial fibrillation requiring treatment (e.g., anti-coagulation and/or antiarrhythmic therapy) within 3 months prior to Screening
4. Recently treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation) within 6 months prior to Screening or plans to have either of these treatments during the study
5. Systolic heart failure with ejection fraction <55% or heart failure symptoms of NYHA Class IV
6. QTcF >480 msec at Screening or Baseline
7. Presence of diseases classified as significant by the Investigator at Screening or Baseline, including the following but not limited to:

   1. Diabetes mellitus requiring treatment
   2. Moderate or severe renal insufficiency or renal insufficiency with estimated glomerular filtration rate <70 mL/min/1.73m2
8. Concomitant use of Disopyramide or Ranolazine within at least 7 days or 5 half-lives (whichever is longer) prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events and their relationship to the investigational product | 12 days

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Tufts Medical Center, Boston, Massachusetts
  - New York University Langone Medical Center, New York, New York
- Poland (2):
  - Independent Public Central Clinical Hospital, Warsaw, Masovian Voivodeship
  - Institute of Cardiology in Warsaw, Warsaw, Masovian Voivodeship
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul